CLINICAL TRIAL: NCT07049419
Title: The Impact of Environmental Controls on Mental Health
Acronym: EC-MH
Status: Completed | Type: Observational
Sponsor: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: AC23092; 23/PR/0917 (Other: London - Harrow Research Ethics Committee)
Record Dates: First submitted 2025-06-19; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Neurologic Disorders
Keywords: Environmental controls; Activities of daily living; Mental health; Self-help devices; Psychological well-being
MeSH Terms: conditions — Nervous System Diseases; Psychological Well-Being

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Environmental control system users: Patients who are eligible for environmental control system users as part of standard clinical care.
  Interventions: Device: Provision of an environmental control system

INTERVENTIONS:
Device: Provision of an environmental control system — Part of standard clinical care for patients referred to the NHS Lothian environmental control service.

SUMMARY:
Within the UK there are over 15 million people who live with at least one long term condition. Of these people, over 4 million suffer from mental health problems.

Environmental control systems are a type of assistive technology that can be controlled by a wide variety of different access methods (e.g. switches) and can assist people with physical disabilities usually with a neurological condition to control various electronic devices in the home environment. The systems are designed to provide independence, removing the requirement to be reliant on other people (for the operation of the controlled devices) and potentially could have a positive effect on mental health and quality of life.

The research question for this study is to determine impact of environmental controls on mental health. It is hypothesised that there will be a positive impact on mental health of the participants. The question above will be answered by collecting questionnaire data pre and post intervention. Participants will be identified by Clinical Scientists working in NHS Lothian's Environmental Control Service (ECS). Participants will be recruited from NHS Lothian and so will be living in the Lothian area. The patient will be contacted following the normal protocol for arranging an environmental control assessment, at which point they will be approached to join the study. Participants will answer questions in their home environment both in person and over the phone.

The end point of the study will be 14 months from the start date (allowing for follow up data to be collected for anyone recruited towards the end of the 12-month recruitment period.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for environmental control system (as per NHS Scotland criteria).
* New user (no previous intervention).
* Neurological condition.
* Cognitive ability to answer the questions and to give consent.

Exclusion Criteria:

* Previous environmental control intervention.
* Patients requiring equipment not supplied by NHS Lothian's ECS (e.g. door interface).
* Patient recently diagnosed (within 6 months).
* Rapidly deteriorating condition.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NHS Lothian patients who have been referred to the Environmental Control Service and are eligible for environmental controls.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
PROMIS Global10 | From enrollment to the end of study period at 8 weeks post installation of the environmental control system.
  A 10 question quality of life outcome measure which can be used to define two separate scores - one for physical health (the PROMIS Global Physical Health score) and one for mental health (the PROMIS Global Mental Health score).
PIADS | From enrollment to the end of study period at 8 weeks post installation of the environmental control system.
  The Psychosocial Impact of Assistive Devices scale (PIADS) was specifically developed for measuring the impact of assistive technology on a participant's psychological well-being, functional independence and quality of life.

SECONDARY OUTCOMES:
Study specific questionnaire | From enrollment to the end of study period at 8 weeks post installation of the environmental control system.
  This includes 3 pre-intervention questions and 6 post-intervention questions. Questions address the use of electronic equipment in the home, how people access their equipment, and their satisfaction and ease of use relating to their environmental control system.

CONTACTS AND LOCATIONS:
Locations (1):
- SMART Centre, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No
IPD is not required to be shared.

DOCUMENTS (1):
  • Study Protocol (2023-10-24): https://cdn.clinicaltrials.gov/large-docs/19/NCT07049419/Prot_000.pdf